CLINICAL TRIAL: NCT01606332
Title: Indwelling Interscalene Nerve Catheters in Surgical Management of Idiopathic Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: OAD Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC001
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single in interscalene block (No Intervention): Single indwelling interscalene block with ropivacaine 0.5% 10ml
- Interscalene block with nerve catheter (Experimental): Interscalene block with ropivacaine 0.5% 10ml and placement of an indwelling nerve catheter with ropivacaine 0.2% @5ml/hr for 24 hours
  Interventions: Procedure: Interscalene block with nerve catheter

INTERVENTIONS:
Procedure: Interscalene block with nerve catheter — Interscalene block with ropivacaine 0.5% 10ml and placement of an indwelling nerve catheter with ropivacaine 0.2% @5ml/hr for 24 hours
  Arms: Interscalene block with nerve catheter

SUMMARY:
In patients who undergo shoulder manipulation for idiopathic adhesive capsulitis, a postoperative indwelling analgesic pain catheter will improve patient outcomes by decreasing shoulder pain and improving range of motion compared to a single-dose interscalene block.

DETAILED DESCRIPTION:
Shoulder manipulation under anesthesia to treat idiopathic adhesive capsulitis is performed only when conservative treatment fails to remedy the condition.

It is common practice to use an interscalene nerve block as anesthesia for this surgical intervention. This randomized prospective study is designed to evaluate the effects of two different anesthesia methods on patient's post-surgical rehabilitation after manipulation. Forty patients scheduled for surgery will be entered into this study. Patients will be randomly assigned to receive a single-doseinterscalene block or a single-dose interscalene block and an indwelling nerve catheter which will provide a continuous infusion of local anesthetic. Patients with the continuous infusion of local anesthetic will receive the additional anesthesia for 24 hours. Patient's range of motion will be evaluated pre-op, intra-op and post-operatively at 10 days, 4,8,16 weeks and 6 months

ELIGIBILITY:
Inclusion Criteria:

* Males and Females over the age of 18 with a diagnosis of idiopathic adhesive capsulitis
* Failed conservative treatment for a minimum of 4 months
* Patient had 3 sequential office visits with no clinical improvement

Exclusion Criteria:

* Adhesive capsulitis following a surgical procedure and/or fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Improvement in shoulder function as demonstrated by increased range of motion | 10 days, 4, 8, 16 weeks and 6 months
  The primary outcome measure will be an improvement in shoulder function as measured by the ASES shoulder score.

SECONDARY OUTCOMES:
Decrease in shoulder pain | 10 days, 4, 8, 16 weeks and 6 months
  The secondary outcome measure will be a reduction in shoulder pain as measured by the VAS pain score.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron A Bare, MD, Principal Investigator — OAD Orthopaedics
Locations (1):
- OAD Orthopaedics, Warrenville, Illinois, United States